CLINICAL TRIAL: NCT07170319
Title: A Phase 1 Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IBI3032 After Multiple Ascending Doses in Participants With Overweight or Obesity
Brief Title: A Study of IBI3032 in Chinese Participants With Overweight or Obesity
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics Technology Limited (Shanghai R&D Center) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI3032T002
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Multiple ascending dose5 of IBI3032 administered orally. (Experimental): Cohort 5 IBI3032
  Interventions: Drug: IBI3032
- Multiple ascending dose1 of placebo administered orally. (Placebo Comparator): Cohort 1 placebo
  Interventions: Drug: placebo
- Multiple ascending dose4 of placebo administered orally. (Placebo Comparator): Cohort 4 placebo
  Interventions: Drug: placebo
- Multiple ascending dose3 of IBI3032 administered orally. (Experimental): Cohort 3 IBI3032
  Interventions: Drug: IBI3032
- Multiple ascending dose4 of IBI3032 administered orally. (Experimental): Cohort 4 IBI3032
  Interventions: Drug: IBI3032
- Multiple ascending dose2 of IBI3032 administered orally. (Experimental): Cohort 2 IBI3032
  Interventions: Drug: IBI3032
- Multiple ascending dose3 of placebo administered orally. (Placebo Comparator): Cohort 3 placebo
  Interventions: Drug: placebo
- Multiple ascending dose5 of placebo administered orally. (Placebo Comparator): Cohort 5 placebo
  Interventions: Drug: placebo
- Multiple ascending dose1 of IBI3032 administered orally. (Experimental): Cohort 1 IBI3032
  Interventions: Drug: IBI3032
- Multiple ascending dose2 of placebo administered orally. (Placebo Comparator): Cohort 2 placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IBI3032 — IBI3032. Method of administration: oral, fasted administration.
  Arms: Multiple ascending dose1 of IBI3032 administered orally.; Multiple ascending dose2 of IBI3032 administered orally.; Multiple ascending dose3 of IBI3032 administered orally.; Multiple ascending dose4 of IBI3032 administered orally.; Multiple ascending dose5 of IBI3032 administered orally.
Drug: placebo — Placebo (without active ingredients). Method of administration: oral, fasted administration.
  Arms: Multiple ascending dose1 of placebo administered orally.; Multiple ascending dose2 of placebo administered orally.; Multiple ascending dose3 of placebo administered orally.; Multiple ascending dose4 of placebo administered orally.; Multiple ascending dose5 of placebo administered orally.

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 1 clinical study evaluating the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of multiple ascending doses of IBI3032 in participants with overweight or obesity. It is a multiple ascending dose study in participants with overweight or obesity during the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females, as determined by medical history
* Have safety laboratory results within normal reference ranges

Exclusion Criteria:

* Have known allergies toIBI3032， glucagon-like peptide-1 (GLP-1) analogs, related compounds
* Abnormal electrocardiogram (ECG) at screening
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-12-24 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One Serious Adverse Event(s) Considered by the Investigator to be Related to Study Drug | Baseline up to Day 43
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module
Number of Participants with More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | Baseline up to Day 43
  A summary of other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Number of Participants with adverse events (AEs) | An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
  Baseline up to Day 43

SECONDARY OUTCOMES:
Under the Serum Concentration-time Curve (AUC) of IBI3032 | Day 1 and Day 28：Predose up to 24 hours postdose. Day 8, Day 15 and Day 22：Predose up to 4 hours postdose.
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
maximum concentration (Cmax) of IBI3032 | Day 1 and Day 28：Predose up to 24 hours postdose. Day 8, Day 15 and Day 22：Predose up to 4 hours postdose.
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
time to maximum concentration (Tmax) of IBI3032 | Day 1 and Day 28：Predose up to 24 hours postdose. Day 8, Day 15 and Day 22：Predose up to 4 hours postdose.
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
clearance (CL) of IBI3032 | Day 1 and Day 28：Predose up to 24 hours postdose. Day 8, Day 15 and Day 22：Predose up to 4 hours postdose.
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
apparent volume of distribution (V) of IBI3032 | Day 1 and Day 28：Predose up to 24 hours postdose. Day 8, Day 15 and Day 22：Predose up to 4 hours postdose.
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
elimination half-life (T1/2) of IBI3032 | Day 1 and Day 28：Predose up to 24 hours postdose. Day 8, Day 15 and Day 22：Predose up to 4 hours postdose.
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- The Frist Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China